CLINICAL TRIAL: NCT06255262
Title: Durvalumab Combined With Surufatinib as Maintenance Therapy in Patients With Advanced Biliary Tract Cancer Whose Disease Did Not Progress After Completion of First-line Durvalumab Combined With Gemcitabine+Cisplatin Treatment
Brief Title: Durvalumab Combined With Surufatinib as Maintenance Therapy in Patients With Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOMESTIC
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Biliary Tract Cancer
Keywords: Maintenance therapy; Durvalumab; Surufatinib
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — surufatinib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab in combination with surufatinib (Experimental): 1. Safety introduction phase (6 cases)
  2. Dose expansion phase (24 cases)
  Interventions: Drug: Surufatinib; Drug: Durvalumab

INTERVENTIONS:
Drug: Surufatinib — (1) Safety introduction phase (6 cases): 250mg, oral, QD,after one cycle of combined treatment, the occurrence of DLT was evaluated: 1) If ≤1person occurs, continue the dose expansion study at that dose level. 2)In the event of DLT> 1, then the dose of surufatinib was adjusted to 200mg，oral，QD,until disease progression or intolerance of toxicity.
  (2) Dose expansion phase (24 cases): RP2D, oral, QD,until disease progression or intolerance of toxicity.
  Other Names: SULANDA; HMPL-012
Drug: Durvalumab — 1500mg, Q4W.iv.every 28 days; until disease progression or intolerance of toxicity.
  Other Names: IMFINZI

SUMMARY:
A Real-World Study of Durvalumab combined with Surufatinib as maintenance therapy in patients with advanced biliary tract cancer whose disease did not progress after completion of first-line Durvalumab combined with Gemcitabine+cisplatin treatment.

DETAILED DESCRIPTION:
This is a single-arm, multicentre real-world study of Durvalumab combined with Surufatinib as maintenance therapy in patients with advanced biliary tract cancer whose disease did not progress after completion of first-line Durvalumab combined with Gemcitabine+cisplatin treatment.The primary purpose of the study is exploring the efficacy and safety of durvalumab in combination with surufatinib for the maintenance therapy of patients with advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years
2. Expected survival is more than 3 months (12 weeks)
3. Patients with unresectable advanced or metastatic BTC confirmed by histopathological and/or cytological examination， including bile duct epithelial cell carcinoma (intrahepatic or extrahepatic), gallbladder
4. Patients received durvalumab plus GemCis as first-line therapy for 4-8 cycles（ Cycles of chemotherapy were determined according to the investigator and safety profile. In addition, durvalumab plus GemCis was considered to be first-line therapy if the patient had received only antineoplastic traditional Chinese medicine or immunomodulatory therapy before treatment ）,without disease progression (i.e., according to the evaluation of RECIST v1.1 CR, PR or SD)
5. At enrollment, World Health Organization (WHO) /ECOG performance status (PS) was 0-1
6. In the first-line treatment at least 1 RECIST 1.1 standard target lesion (TL)
7. Organs and bone marrow are sufficiently functional, defined as follows:

   Hemoglobin ≥7g/dL Absolute neutrophil count ≥1.5 × 109/L The platelet count was ≥ 90 × 109/L Serum bilirubin ≤2.0 × upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be 2.5 × ULN or less. For patients with liver metastases, ALT and AST should be ≤5 × ULN Creatinine clearance, calculated by means of the Cockcroft-Gault (based on actual body weight) formula or the 24-hour urinary creatinine clearance assay, should be greater than 50 mL /min
8. Weight: > 30kg
9. Female subjects promised to be nonpregnant before enrollment, had to be nonlactating, and agreed to use highly effective contraception for the duration of the study
10. Male patients who had sex with a female partner of potential pregnancy had to use an acceptable method of contraception from screening through the duration of the study and the drug washout period to prevent their partner from becoming pregnant
11. Patients voluntarily participated in the trial, signed informed consent, and complied with the agreement, including receiving treatment, regular visits and examinations, and follow-up.

Exclusion Criteria:

1. Carcinoma of ampulla
2. Any evidence of disease, as judged by the investigator（such as severe or uncontrolled systemic disease, including hypertension that is not controlled by drugs, active bleeding disease, active infection, active ILD/ interstitial lung disease, severe chronic gastrointestinal disease related to diarrhea, mental illness/social conditions）, or a history of allogeneic transplantation that was deemed by the investigator to be inappropriate for study participation or to interfere with adherence to the study protocol
3. Active or previously documented autoimmune or inflammatory disease, these include inflammatory bowel diseases [such as colitis or Crohn's disease], diverticulitis [except diverticulosis], systemic lupus erythematosus, sarcoid syndrome, Wegener syndrome [granulomatosis with polyangiitis], Graves disease, rheumatoid arthritis, hypophysitis and uveitis. Exceptions to this criterion are made in the following cases:

   Subjects with vitiligo or alopecia ubjects with hypothyroidism (e.g., after Hashimoto's syndrome) whose condition is stable with hormone-replacement therapy Subjects with any chronic skin disease who did not require systemic treatment Subjects who had not had active disease within the previous 5 years could be enrolled, but only after consultation with a study physician Subjects with celiac disease that could be controlled by diet alone Subjects with ≥ grade 2 lymphopenia will be evaluated on a case-by-case basis after consultation a graduate physician.
4. A history of other primary malignancies, except for:Malignancies treated with curative treatment, known no active disease for more than 5 years before the first study intervention, and low potential recurrence；Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or lentigo maligna that has received potentially curative treatment；Or carcinoma in situ that has been adequately treated without evidence of disease
5. History of meningeal carcinomatosis
6. A history of active primary immunodeficiency
7. Active infections, including tuberculosis (clinical assessment, including the clinical history, physical examination and imaging results, and on the basis of the local operation of tuberculosis examination), or human immunodeficiency virus (HIV 1/2 antibody positive)
8. Other approved or investigational antiangiogenic tyrosine kinase inhibitors or monoclonal antibodies were received before the initiation of study treatment
9. Caused by past anti-tumor treatment for toxic effects (CTCAE>Grade 2), except for alopecia and vitiligo Subjects with ≥ grade 2 neurological disease will be evaluated on a case-by-case basis after consultation with the study physician Subjects who had an unreasonable expectation of worsening irreversible toxicity from treatment with durvalumab had to consult a study physician before they could be enrolled
10. Existing medical conditions or history of brain metastases or spinal cord compression (including asymptomatic and adequately treated disease)
11. Known allergies or hypersensitivity reactions to any of the study intervention treatments or any of the study intervention treatment excipients
12. Any medical, biologic, or hormonal therapy for cancer that was not permitted in the protocol was used concomitantly. At the same time use hormone therapy of tumor related diseases (such as hormone replacement therapy) is acceptable
13. Patients had received live attenuated vaccine within 30 days before the first dose of the study intervention. During the study intervention therapy and the last up to 30 days after the drug into the group of patients are not allowed to accept live vaccine inoculation
14. Major surgical procedure (investigator-defined) within 28 days before the first dose
15. Participants were enrolled in another clinical trial within 30 days before enrollment and received the investigational drug and any concomitant therapy containing the investigational drug
16. Any of the following events occurred within 6 months before enrollment: myocardial infarction, severe/unstable angina, coronary/peripheral-artery bypass grafting, congestive heart failure in NYHA class III or IV, stroke, or transient ischemic attack
17. Any serious acute or chronic medical condition that would prevent the patient from participating in the study or affect the interpretation of the study results
18. Pregnant or lactating women. Pregnancy status was known before enrollment
19. Patients of childbearing age (male/female) who do not agree to use an accepted effective method of contraception during the study treatment and for at least 6 months after the completion of the study treatment
20. If urine routine test showed urine protein ≥2+ and 24-hour urine protein >1.0g
21. Other strong inducers or inhibitors of CYP3A4 were taken within 2 weeks before the first study dose
22. Othere conditions that the investigator thought should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival 1 (PFS1) | 2 years
  PFS1 defined as the time from the initiation of first-line treatment to tumor progression or death.

SECONDARY OUTCOMES:
Safety(number and degree of adverse events) | 2 years
  Safety and tolerance assessment will be conducted according to AE with CTCAE grade ≥3, AESI, ADR, AE, imAE and SAE.
Progression-free survival 2 (PFS2) | 2 years
  Defined as the time from the initiation of maintenance therapy to tumor progression or death.
1-year survival rate（OS12） | 2 years
  Defined as the KM estimate of OS at 12 months after the first dose of first-line therapy, OS12 and 95% CI will be summarized using the Kaplan-Meier method.
Objective Response Rate(ORR,investigator-assessed RECIST 1.1/mRECIST) | 2 years
  Defined as the number of patients (%) with at least one CR or PR visit response since first-line therapy. ORR assessments will include data obtained before progression or before the last evaluable assessment in the absence of progression.ORR will be summarized with the use of the Clopper-Pearson (exact) method and expressed as percentages with 95% confidence intervals.
Disease Control Rate(DCR) | 2 years
  Defined as the best objective response rate of CR, PR, or SD according to RECIST 1.1/ mRECIST criteria. The DCR will be analyzed in the same way as ORR.
Duration of Response(DoR) | 2 years
  Defined as the date of first documented response to disease progression or occurrence of death with or without disease progression (i.e., PFS event or censoring date - date of first response +1). The end date of disease response should coincide with the date of progression or death from any cause used for the PFS endpoint. The time to first response was defined as the follow-up date of the first assessment of CR or PR since the initiation of first-line therapy.
Overall Survival(OS) | 2 years
  Defined as the time from the first dose of first-line therapy to death, irrespective of the actual cause of death of the subject. OS for subjects who were still alive at the time of data analysis or lost to follow-up was censored at the last recording date, that is, subjects known to be alive at or before the data analysis cutoff date.

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, PhD, Principal Investigator — First Hospital of China Medical University; Xiujuan Qu, PhD, Principal Investigator — First Hospital of China Medical University
Locations (4):
- China (4):
  - Anshan Cancer Hospital, Anshan, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning
  - Shenyang Fifth People's Hospital, Shenyang, Liaoning